CLINICAL TRIAL: NCT04894565
Title: Effectiveness of Home-based and Early Institutional Physiotherapy Program for Breast Cancer Women Following Surgery: A Pilot Clinical Trial
Brief Title: Physiotherapy Program for Breast Cancer Women Following Surgery: A Pilot Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Hussam Sakkijha, Principal Investigator, King Fahad Medical City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-115
Record Dates: First submitted 2021-05-06; First posted 2021-05-20 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Consecutive women with breast cancer who underwent breast cancer surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): effect of rehabilitation program in the intervention arm
  Interventions: Procedure: rehabilitation

INTERVENTIONS:
Procedure: rehabilitation — physical therapy 24 hrs after surgery

SUMMARY:
pilot study on physical therapy in women with breast cancer immediately following surgery

DETAILED DESCRIPTION:
A pilot, single-arm non-randomized clinical trial was conducted between the period September 2018 and June 2019 on a convenient sample of BC women. Primary study outcomes were pain, disabilities of the Arm, Shoulder, and Hand (DASH), handgrip strength, and quality of life (QoL). The secondary outcome was to assess the feasibility of this pilot study. All outcomes were recorded at three time- intervals (T0=day 1 post-operation), (T1=day 30), and (T1=day 90) under standardized conditions. The interventions were delivered by the physiotherapist early within 24 hours post-operatively, T1, and T2. In addition, home-based exercise was provided with written instructions during hospitalization with rehearsal sessions to ensure the patient's understanding and compliance

ELIGIBILITY:
Inclusion Criteria:

* women with breast cancer who require surgical resection

Exclusion Criteria:

* in ability to undergo 3 months of physical therapy program

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women with breat cancer
Enrollment: 23 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Shoulder/Arm Pain | The measurements of the study outcomes took place at three time- intervals (T0=day 1 post-operation), (T1=day 30), and (T1=day 90).
  Pain in the shoulder/arm was assessed using the visual analogue scale (VAS) with a scoring system of 0-10 (0 = no pain; 1-3; mild pain, 4-6; moderate pain, 7-10 severe pain)
Shoulder mobility | The measurements of the study outcomes took place at three time- intervals (T0=day 1 post-operation), (T1=day 30), and (T1=day 90).
  Shoulder mobility (flexion [0-180°], abduction [0-180°]) was measured by using a digital inclinometer under standardized conditions. Patients were maintained in a seated position for all movements to minimize compensatory movements of the trunk.
Disabilities in daily life | The measurements of the study outcomes took place at three time- intervals (T0=day 1 post-operation), (T1=day 30), and (T1=day 90).
  by using Quick DASH scale (Disabilities of the Arm, Shoulder, and Hand) questionnaire. The Quick DASH consists of 11 items that allow for cumulative and multiple assessments of a patient over time, and each item has 5 response options. According to the Quick DASH scale scoring system, the scale scores are calculated and ranging from 0 (no functional disability) to 100 (most severe disability)
Handgrip strength | The measurements of the study outcomes took place at three time- intervals (T0=day 1 post-operation), (T1=day 30), and (T1=day 90).
  measured while the patient stabilized in a seated position with the elbow in 90 degrees of flexion and squeezes three times the dynamometer with each hand.
Quality of Life (QoL) | The measurements of the study outcomes took place at three time- intervals (T0=day 1 post-operation), (T1=day 30), and (T1=day 90).
  Patients' QoL was assessed by using the Functional Assessment of Cancer Therapy-General (FACT-G) scale. FACT-G (version-4) is a validated, self-reported multi-dimensional, 27-items questionnaire measuring QoL for breast cancer patients with 1 4-points Likert scale (0-108). The FACT-G comprises of 4-subscales: Physical Well-being (PWB: 7-items; score range 0 to 28), Social Well-being (SWB: 7-items; score range 0 to 28), Emotional Well-being (EWB: 6-items; score range 0 to 24), Functional Well-being (FWB: 7-items; score range 0 to 28)

SECONDARY OUTCOMES:
Establishing firmly study feasibility | 3 months
  Assess for clinical effect size (ES) worth investigation, sample recruitment strategy, adherence to study protocol, and adverse events in preparation to conduct a larger definitive study.

CONTACTS AND LOCATIONS:
Overall Officials: Noura Binsaad, MD, Principal Investigator — Consultant
Locations (1):
- KFMC, Riyadh, Saudi Arabia